CLINICAL TRIAL: NCT03423914
Title: Efficacy of Expressive Writing in Mothers of Hospitalized Preterm Infants
Brief Title: Efficacy of Expressive Writing in Mothers of Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Industrial de Santander (Other)
Responsible Party: Principal Investigator, Martha Isabel Camargo, Associate Nursing Professor, Universidad Industrial de Santander
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 10620
Record Dates: First submitted 2018-01-18; First posted 2018-02-06 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Premature Infant; Mothers
Keywords: writing; postraumatic stress; coping
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Mixed study, where the quantitative and qualitative. From the quantitative is an experimental study type controlled clinical trial. From the qualitative it will be interpretive phenomenological
Who Masked: Participant, Care Provider
Masking Description: random allocation of the mother to the control or intervention group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Writing Intervention Group (Experimental): Expressive writing The participant will write four days about her deepest thoughts and feelings in relation to the experience of hospitalization of the premature newborn and how this experience is related to your current life and to your future.
  Interventions: Behavioral: Expressive writing
- Control Group (Active Comparator): Only Writing The participants will write about situations not related to the subjective human experience of their preterm birth, but about general aspects.
  Interventions: Other: Only Writing

INTERVENTIONS:
Behavioral: Expressive writing — The emotional or expressive writing therapy developed by James Pennebaker has been used as a method of self-understanding in people with high levels of stress, chronic diseases, sexual and physical abuse, natural disasters and job loss, among others. Expressive writing allows and implies revealing the deepest thoughts and feelings of the person about a stressful or traumatic event in life translate emotions into words, and with that, reduce mental stress (decrease in levels of depression, stress and anxiety), strengthen self-esteem and even strengthen the immune system
  Arms: Writing Intervention Group
Other: Only Writing — Participants write about knowledge related to infant care during four days
  Arms: Control Group

SUMMARY:
Premature birth can lead the mother to lose control of herself, and be a contributor to the psychological stress experienced due to the sudden breakdown of the interaction with her infant because of hospitalization in a neonatal care unit. This is a mixed method study, the aim is establish the effectiveness of expressive writing in the experience of mothers of hospitalized preterm infants. The intervention Expressive writing therapy could contribute to reduce the level of stress and anxiety, improving coping and the mother's interaction with her infant.

DETAILED DESCRIPTION:
Background: The literature has shown the application of expressive writing therapy after traumatic events, and the measurement of its impact on people´s health through the application of quantitative instruments. However, no studies have been carried out in which this therapeutic activity has been measured with quantitative methods and at the same moment, to measure the experience using qualitative analysis that allows to understand in depth the human experience. Expressive writing therapy could contribute to reducing the level of stress and anxiety, improving coping and the interaction of the mother with her premature newborn (PNTBs). In this sense, it is necessary to have a scientific research in this area, from a qualitative-quantitative approach allows demonstrating the reach of positive effects in the emotional health status of mothers with PTNBs hospitalized in a neonatal care unit (NICU).

General purpose: To establish the effectiveness of expressive writing in the experience of mothers of hospitalized preterm infants.

Specific objectives:

* Establish the coping capacity of the mothers of the premature Infants before and after the intervention.
* Determine the level of post-traumatic stress of the mothers of the premature Infants before and after the intervention.
* Establish the performance of the maternal role of the mothers of the premature Infants before and after the intervention.
* Describe how mothers of RNPT experience the experience of having their child hospitalized
* Understand the meaning of the mother's experience in the transition to the maternal role of a premature

Design: Mixed study, where the quantitative and qualitative method is used. Which allows to combine the two paradigms to approach in a more integral way to the research problematic. In this sense, the research will be strengthened, to be able to incorporate data from the writing of the participants to give greater meaning to the numerical data. From the quantitative is an experimental study type controlled clinical trial. From the qualitative, it will be interpretative phenomenological; philosophical methodology that allows to discover and understand the meaning of human experience around a phenomenon.

For the measurement of the results before and after the intervention, the Nursing Outcome -NOC: Performance of the maternal role (2211) will be applied to both groups. In the experimental group the Nursing Intervention will be applied- NIC: Journalist (4740)

Population of study: Mothers with premature newborns hospitalized in the neonatal care unit at third level Hospital in Bucaramanga, Colombia.

Sample Size: For the quantitative design, the sample size was calculated taking into account, according to previous studies the change of 2.5 in the PST scale to achieve a decrease in the levels of post-traumatic stress. This study will randomly allocate 60 premature infant´s mothers, 30 for each group, with a power of 80% and an alpha of 0.05. For the qualitative design, convenience sampling will be taken into account from the writings made by the mothers of the intervention group.

Inclusion Criteria: Mothers with:

* Age of 14 or more years old
* Preterm newborns with a gestational age of less than 34 weeks
* Preterm newborns who are hospitalized in the NICU of the Third level Hospital of Santander
* Preterm newborns alive at the time of assignment to the control group or intervention group
* The time of hospitalization of the newborn must be at least one week in the hospital institution.
* Nursing Diagnosis Readiness of enhanced parenting (00164)

Exclusion Criteria:

Mother with

* Limitations like as hearing, motor and / or mental disability - measured through the minimental test.
* Consumption of psychoactive substances
* Mothers who can not read or write
* Newborns with a confirmed diagnosis of severe diseases as a congenital malformations.

Instruments: Coping level scale, Perinatal posttraumatic stress scale, maternal role performance scale, Minimental test

ELIGIBILITY:
Inclusion Criteria:

Mothers with:

* Age of 14 or more years old
* Preterm newborns with a gestational age of less than 34 weeks
* Preterm newborns who are hospitalized in the NICU of the third level Hospital of Santander
* Preterm newborns alive at the time of assignment to the control group or intervention group
* The time of hospitalization of the newborn must be at least one week at the hospital.
* Nursing Diagnosis Readiness for enhanced parenting (00164)

Exclusion Criteria:

* Limitations as hearing, motor and / or mental disability measured through the minimenta test.
* Active consumption of psychoactive substances
* Mothers who can not read or write,
* Mothers of newborns with a confirmed diagnosis of severe diseases like congenital malformations.

Ages: 14 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Posttraumatic stress | fifth day
  Decreased of stress in mothers. It will be measure using the Postnatal Perinatal Stress Scale, a 14-item questionnaire that examines maternal perinatal post-traumatic stress symptoms specific to childbirth. The scores range between 0 and 14; but a score of 6 would qualify for a diagnosis of PTSD

SECONDARY OUTCOMES:
Coping and adaptation | fifth day
  Improve coping and adaptacion in mothers of premature infants. Level of coping scale: It is the instrument that allows the identification of coping and adaptation strategies used by people to face difficult situations. It is a measurement scale that contains 33 indicators each with 4 Likert type response options from never to always. Each item is a short phrase that describes how a person responds when they have a critical or difficult situation

CONTACTS AND LOCATIONS:
Overall Officials: Martha Camargo, RN-MsC, Principal Investigator — Associate Professor
Locations (1):
- Hospital Universitario de Santander, Bucaramanga, International, Colombia

IPD SHARING:
Plan to Share IPD: Undecided
The publication of the results of this study will be carried out in an indexed journal and in scientific events.

REFERENCES:
- [Background] Hawes K, McGowan E, O'Donnell M, Tucker R, Vohr B. Social Emotional Factors Increase Risk of Postpartum Depression in Mothers of Preterm Infants. J Pediatr. 2016 Dec;179:61-67. doi: 10.1016/j.jpeds.2016.07.008. Epub 2016 Aug 5. PMID 27502105
- [Background] Aftyka A, Rybojad B, Rosa W, Wrobel A, Karakula-Juchnowicz H. Risk factors for the development of post-traumatic stress disorder and coping strategies in mothers and fathers following infant hospitalisation in the neonatal intensive care unit. J Clin Nurs. 2017 Dec;26(23-24):4436-4445. doi: 10.1111/jocn.13773. Epub 2017 Apr 20. PMID 28231614
- [Background] Yang YY, He HG, Lee SY, Holroyd E, Shorey S, Koh SSL. Perceptions of Parents With Preterm Infants Hospitalized in Singaporean Neonatal Intensive Care Unit. J Perinat Neonatal Nurs. 2017 Jul/Sep;31(3):263-273. doi: 10.1097/JPN.0000000000000239. PMID 28234668
- [Background] Wormald F, Tapia JL, Torres G, Canepa P, Gonzalez MA, Rodriguez D, Escobar M, Reyes B, Capelli C, Menendez L, Delgado P, Treuer S, Ramirez R, Borja N, Dominguez A; Neocosur Neonatal Network (Red Neonatal Neocosur). Stress in parents of very low birth weight preterm infants hospitalized in neonatal intensive care units. A multicenter study. Arch Argent Pediatr. 2015 Aug;113(4):303-9. doi: 10.5546/aap.2015.eng.303. English, Spanish. PMID 26172004